CLINICAL TRIAL: NCT06599697
Title: The MIGHT Trial - An Exploratory Clinical Trial of Intravenous Immunoglobulin (IVIG) in Anti-3-Hydroxy-3-Methylglutaryl-CoA Reductase (HMGCR) Immune Mediated Necrotizing Myopathy (IMNM)
Brief Title: The MIGHT Trial - An Exploratory Clinical Trial of IVIG in Anti-HMGCR Immune Mediated Necrotizing Myopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Octapharma USA, Inc. (Unknown); CSI Pharmacy (Unknown)
Responsible Party: Principal Investigator, James Andrews, Assistant Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300013467; 1R21AR083566-01A1 (NIH)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anti-3-hydroxy-3-methylglutaryl-CoA Reductase (HMGCR) Immune-Mediated Necrotizing Myopathy

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, double blinded phase 2 exploratory clinical trial of intravenously administered pooled human immunoglobulin (IVIG) in anti-3-hydroxy-3-methylglutaryl-CoA reductase (HMGCR) immune mediated necrotizing myopathy (IMNM). Planned enrollment is 12 individuals with active anti-HMGCR IMNM meeting inclusion and exclusion criteria. Enrolled participants will be randomized 1:1 to receive either IVIG 2g/kg or placebo (0.9% sodium chloride at equivalent volume) at weeks 0, 4, and 8. The 2g/kg q4 weeks regimen of IVIG was chosen based on the investigators' clinical experience and prior studies. The primary endpoints will be assessed at week 12. After the randomized phase of the trial, all participants will be offered an open-label extension to receive IVIG at weeks 12, 16, and 20.
Who Masked: Participant, Investigator
Masking Description: Using an online randomization tool (e.g. REDCap), 12 total participants will be randomized 1:1 in blocks of 4 to receive either intravenously administered pooled human immunoglobulin (IVIG) 2g/kg every 4 weeks or placebo (0.9% sodium chloride solution at equivalent volume to corresponding IVIG weight-based dose). The home infusion research pharmacy (CSI Pharmacy) will assign treatment status using the randomization tool and will prepare IVIG or placebo for home infusion nursing staff in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenously Administered Pooled Human Immunoglobulin (IVIG) (Experimental): Participants will receive intravenously administered pooled human immunoglobulin (IVIG) 2g/kg every 4 weeks for 24 weeks.
  Interventions: Biological: Intravenously administered pooled human immunoglobulin (IVIG)
- Placebo (No Intervention): Participants will receive an infusion of 0.9% sodium chloride solution every 4 weeks for 16 weeks at equivalent volume to corresponding IVIG weight-based dose.

INTERVENTIONS:
Biological: Intravenously administered pooled human immunoglobulin (IVIG) — IVIG 2g/kg every 4 weeks for 12 weeks (3 doses)
  Other Names: Octagram -Immune Globulin Intravenous (Human)
  Arms: Intravenously Administered Pooled Human Immunoglobulin (IVIG)

SUMMARY:
This is a randomized, placebo-controlled, double blinded phase 2 exploratory clinical trial of intravenously administered pooled human immunoglobulin (IVIG) in anti-3-hydroxy-3-methylglutaryl-CoA reductase (HMGCR) immune mediated necrotizing myopathy (IMNM). Planned enrollment is 12 individuals with active anti-HMGCR IMNM meeting inclusion and exclusion criteria. Assuming 20% drop-out, the investigators anticipate 10 participants will complete all study assessments. Enrolled participants will be randomized 1:1 to either IVIG 2g/kg or placebo (0.9% sodium chloride at equivalent volume) at weeks 0, 4, and 8. The primary efficacy and co-primary safety and tolerability endpoints will be assessed at week 12. After the randomized phase of the trial, all participants will be offered to continue on to an open-label extension phase in which participants will receive IVIG at weeks 12, 16, and 20. Participants will then return at week 24 for a final non-infusion visit to reassess safety, tolerability, and efficacy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Anti-HMGCR antibody positive
* MMT-8 score < 142 (range 0-160)
* Serum CK > 5x upper limit of normal
* Anti-HMGCR IMNM disease duration < 36 months at screening
* No moderate or severe respiratory or swallowing dysfunction due to anti-HMGCR IMNM at screening
* No history of dermatomyositis rash
* Must reside in a state with a participating research site

Exclusion Criteria:

* Oral glucocorticoid (GC) daily dose > 15mg at screening
* Change in oral GC dose < 2 weeks prior to screening
* Prior IVIG treatment for anti-HMGCR IMNM

  ->1 oral conventional synthetic DMARD (e.g. methotrexate, mycophenolate mofetil, azathioprine) use at screening
* Change in concomitant DMARD dose < 4 weeks prior to screening
* Rituximab < 6 months prior to screening
* Plasma exchange, cyclophosphamide, or biologic immunosuppressive medication < 3 months prior to screening
* Use of statin medication at screening
* History of anaphylactic reaction to IVIG
* History of angina pectoris, myocardial infarction, transient ischemic attack, or stroke < 12 months prior to screening
* Females of child-bearing potential who are pregnant, breastfeeding, or are unwilling to practice a highly effective method of contraception during the study
* Wells Criteria for DVT score of 2 or more at screening
* Wells Criteria for PE score of 4 or more at screening
* Weight >120kg
* History of cancer (excluding non-melanomatous skin cancer) < 5 years prior to screening
* History of pulmonary embolism or deep venous thromboembolism < 3 years prior to screening
* History of hyperviscosity or hypercoagulable state
* Currently receiving anti-coagulation therapy (vitamin K antagonists, non-vitamin K oral anticoagulants [e.g. dabigatran, rivaroxaban, apixaban], parenteral anticoagulants [e.g. fondaparinux]. Note that oral anti-platelet agents are allowed (e.g. aspirin, clopidogrel, ticlopidine).
* Glomerular filtration rate (GFR) <60mL/min at the time of screening
* Any medical condition which, in the investigator's judgment, makes participation in the clinical trial unadvisable or which would interfere with evaluation of the study treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change in serum creatine kinase (CK) | Week 0 to 12
  Primary Efficacy Outcome

CONTACTS AND LOCATIONS:
Overall Officials: James Andrews, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided